CLINICAL TRIAL: NCT00269438
Title: Phase 3 Study to Establish the Efficacy and Safety of a New Tablet Formulation and Dosing Regimen of Balsalazide Disodium Dosed Twice Daily in Achieving Clinical Improvement in Subjects With Mildly to Moderately Active Ulcerative Colitis After 8 Weeks of Therapy
Brief Title: New Tablet Formulation and Dosing Regimen of Balsalazide Disodium in Mildly to Moderately Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BZUC3002
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; Enema; Suppositories; Adrenal Cortex Hormones

INTERVENTIONS:
Drug: 5 ASA, enemas, suppositories, corticosteroids

SUMMARY:
The purpose of this study is to establish the efficacy and safety of a new tablet formulation and dosing regimen of balsalazide disodium dosed twice daily in achieving clinical improvement in subjects with mildly to moderately active ulcerative colitis after 8 weeks of therapy.

DETAILED DESCRIPTION:
The primary efficacy endpoint is the proportion of subjects that achieve clinical improvement and improvement in the rectal bleeding subscale of the MMDAI at the end of eight weeks of therapy, where clinical improvement is defined as a greater than or equal to 3 point improvement from baseline in the MMDAI.

The secondary endpoints are as follows:

1. The change from baseline over the duration of treatment in total MMDAI score and in the individual MMDAI subscales.
2. The change from baseline to Weeks 1, 2, 4 and 8 in total MMDAI score and in each individual MMDAI subscale (endoscopy/sigmoidoscopy at Weeks 2 and 8 only).
3. The proportion of subjects with treatment failure, defined as withdrawal due to significant disease progression or lack of significant improvement, as determined by the Investigator.
4. The proportion of subjects with mucosal healing at Weeks 2 and 8, where mucosal healing is defined as an endoscopy/sigmoidoscopy score of 0 or 1
5. The proportion of subjects achieving complete remission at Week 2 and Week 8, where complete remission is defined as a MMDAI score of less than or equal to 1.
6. The proportion of subjects with improvement from baseline to Weeks 1, 2, 4 and 8 in total MMDAI score and in each individual MMDAI subscale (endoscopy/sigmoidoscopy at Weeks 2 and 8 only).
7. Change from baseline to Weeks 1, 2, 4 and 8 in diarrhea, abdominal discomfort, and subjective sense of well being, as recorded in the subjects' diaries.
8. The proportion of subjects achieving clinical remission at Weeks 1, 2, 4 and 8, where clinical remission is defined as a score of 0 for rectal bleeding and a combined score of less than or equal to 2 for bowel frequency and physician assessment using the MMDAI.
9. Time to clinical remission, where clinical remission is defined as in secondary endpoint number eight.

Safety endpoints are as follows:

* incidence of treatment-emergent AEs grouped by body system and evaluated by treatment group;
* changes from baseline in clinical laboratory parameters at each treatment visit by treatment group; and
* changes from baseline in vital sign measurements at each treatment visit by treatment group.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
2. Subject is a male or, if the subject is female, she is eligible to enter if she is of:

   Non-childbearing potential (i.e. physiologically incapable of becoming pregnant, including any female who has undergone sterilization [hysterectomy or bilateral tubal ligation] or is post-menopausal. For purposes of this study, postmenopausal is defined as 1 year without menses);

   OR,

   Childbearing potential, has a negative serum pregnancy test at screen and, if heterosexually active, agrees to one of the following:
   * Double barrier method of contraception, specifically, use of a condom and spermicide, for 1 week prior to study drug administration, throughout the 8 week Treatment Phase.
   * Oral contraceptives administered for at least 2 monthly cycles prior to study drug administration during all 6 months of study drug administration and administered for 1 monthly cycle following completion of the study.
   * An intrauterine device (IUD), inserted by a qualified clinician, with published data showing that the lowest expected failure rate is less than or equal to 1% per year (not all IUDs meet this criterion).
   * Medroxyprogesterone acetate (DEPO-PROVERA) administered for a minimum of 1 monthly cycle prior to the study drug administration, during all 6 months of study drug administration, and administered for 1 monthly cycle following study completion. Norelgestromin/ ethinyl estradiol transdermal system (Ortho Evra patch) administered for at least 2 monthly cycles prior to study drug administration and administered for 2 monthly cycles following study completion
   * Partner has undergone vasectomy and subject is in a monogamous relationship. The investigator is responsible for determining whether the subject is using appropriate birth control for study participation.
   * Subject is greater than or equal to 18 years of age.
   * Subjects with mildly to moderately active ulcerative colitis experiencing symptoms of an acute flare within the past 4 weeks.
3. Subject has not taken more than 2.4 grams of mesalamine or equivalent for a continuous period of 4 weeks preceding the screening visit
4. Subjects must have a baseline Modified Mayo Disease Activity Index (MMDAI) score between 6 and 10, inclusive. Additionally, subjects must score greater than or equal to 2 on Bleeding and greater than or equal to 2 on Endoscopy/Sigmoidoscopy.
5. Subject is capable and willing to comply with all study procedures.
6. Disease extends at least 20 cm from the rectum on screening sigmoidoscopy.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply (Note: Development of any of the following exclusion criteria on-study will be considered a basis for subject discontinuation.):

1. Subject has a significant medical, including psychiatric, condition which in the opinion of the investigator precludes participation in the study.
2. Subject has a history of allergy or intolerance to aspirin, mesalamine, or other salicylates.
3. Subject has recently (within the past 30 days) failed therapy with balsalazide disodium
4. Subject has received immunosuppressive therapy (e.g. azothioprine, 6 mercaptopurine) within 30 days, or corticosteroids (oral, intravenous [IV] or topical rectal) within 30 days prior to screening.
5. Subject has received intra-rectal aminosalicylates within 14 days of screening.
6. Subject has had any prior bowel surgery, excepting appendectomy.
7. Subject has participated in an investigational drug or device study within the 30 days prior to study screening, with the exception of Salix protocols 3003 & 3004 entitled: "A multicenter, randomized, double-blind, placebo controlled trial to evaluate the use of mesalamine pellet formulation 1.5G QD to maintain remission from mildly to moderate ulcerative colitis."
8. Subject is pregnant or at risk of pregnancy, or is lactating (female subjects only).
9. Subject shows evidence of current excessive alcohol consumption or drug dependence.
10. Subject has a history of human immunodeficiency virus (HIV) or hepatitis (B and C).
11. Subject has other infectious, ischemic, or immunologic diseases with GI involvement.
12. Subject has twice the upper limit of normal (ULN) for any of the following LFTs: alanine aminotransferase (ALT/SGPT), aspartate aminotransferase (AST/SGOT), alkaline phosphatase, or total bilirubin (except isolated elevation of unconjugated bilirubin).
13. Subject has uncontrolled, clinically significant renal disease manifested by 1.5 × ULN of serum creatinine or blood urea nitrogen (BUN) levels.
14. Subject has calculated creatinine clearance level of less than or equal to 60 mL/min.
15. Subject has unstable cardiovascular, coagulopathy or pulmonary disease.
16. Subject has active malignancy within the last 5 years, except basal cell carcinoma of the skin, or if female, in situ cervical carcinoma that has been surgically excised.
17. Subject has any condition or circumstance that would, in the opinion of the investigator, prevent completion of the study or interfere with analysis of study results, including history of noncompliance with treatments or visits.
18. Subject has sclerosing cholangitis.
19. Subject has positive stool culture for ovum and parasites (O and P) or C. difficile.
20. Subject has been treated with infliximab, cyclosporine, natalizumab, or methotrexate for ulcerative colitis within the last 30 days prior to screening.
21. Regular use of NSAIDS except cardioprotective ASA (i.e., less than or equal to 162 mg ASA per day).
22. Subject has received cell-depleting therapies such as the Adacolumn.
23. Subject requires antidiarrheal therapy during screening.
24. Subject has clinical or radiographic findings suggestive of serious UC complications such as toxic megacolon or colonic perforation.

Females of Reproductive Potential:

If a female subject becomes pregnant while on this study, the study drug will be discontinued immediately and the subject followed until the outcome of the pregnancy is known. If a pregnancy occurs, it will be reported in the same manner as an unexpected AE using the guidelines provided in Section 6.4.1.9.

Premature Subject Discontinuation:

A subject may be discontinued from the study for the following medical or administrative reasons:

* Occurrence of an AE, which in the judgment of the investigator suggests an unacceptable risk to the subject (The investigator will follow the subject until satisfactory resolution of the AE or the AE is determined to be stable);
* Development on-study of any condition which, in the opinion of the investigator or the study sponsor, places the subject at an unacceptable medical risk if he/she continues;
* Pregnancy;
* Subject request;
* Institution of additional medical (rescue) therapy for UC. The investigator may discontinue individual subjects from the study at any time. Subjects will be encouraged to complete the study; however they may voluntarily withdraw at any time. The investigator must provide written documentation of the reason for discontinuation on the CRF. Regardless of the reason for withdrawal, all subjects will be asked to undergo an end of therapy evaluation. Every attempt will be made to obtain all the end of study assessments, including all of the subscales of the MMDAI (i.e., bowel frequency, bleeding, physician's assessment, and endoscopy/sigmoidoscopy score).

Subjects who withdraw or are withdrawn will not be replaced under this protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225
Dates: Start 2005-12; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects that achieve clinical improvement and improvement in the rectal bleeding subscale of the MMDAI at the end of eight weeks of therapy, where clinical improvement is defined as a >3 point improvement from baseline in the MMDAI.

SECONDARY OUTCOMES:
The change from baseline over the duration of treatment in total MMDAI score and in the individual MMDAI subscales.

CONTACTS AND LOCATIONS:
Locations (66):
- United States (66):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - Spring Memorial Hospital, Mobile, Alabama
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Lovelace Scientific Resources, Beverly Hills, California
  - Digestive Liver Disease Specialists, Medical Group, Garden Grove, California
  - Therapeutic Research Institute of Orange County, Laguna Hills, California
  - Long Beach VA Medical Center, Long Beach, California
  - Facey Medical Group, Mission Hills, California
  - Community Clinical Trials, Orange, California
  - Rider Research Group, San Francisco, California
  - John Jolley, M.D., San Rafael, California
  - Lovelace Scientific Resources, Santa Ana, California
  - Santa Barbara Clinical Research, Santa Barbara, California
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Stamford Therapeutic Consortium, Stamford, Connecticut
  - Medical Research Unlimited, Hialeah, Florida
  - Mark Lamet, M.D., Hollywood, Florida
  - Southern Clinical Research Consultants, Hollywood, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - Venture Research Institute, LLC, North Miami Beach, Florida
  - Advanced Gastroenterology Associates, Palm Harbor, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Advent Clinical Research, Sarasota, Florida
  - Clinical Research of Tampa Bay, Inc., Spring Hill, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Gary Richter, M.D., Atlanta, Georgia
  - The Atlanta Center for Gastroenterology, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Northwest Gastroenterologists S.C., Arlington Heights, Illinois
  - University Digestive Health Center, Oak Forest, Illinois
  - Covenent Clinic, Waterloo, Iowa
  - Digestive Health Center, Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - Digestive Health Center of Louisiana, Baton Rouge, Louisiana
  - Woodholme Gastroenterology Associates, PA, Baltimore, Maryland
  - Sinai Medical Office Building, Baltimore, Maryland
  - Mid Atlantic Medical Research Centers, Hollywood, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Kansas City, Missouri
  - Center for Digestive & Liver Diseases, Mexico, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Central Jersey Primary Care Inc., Elizabeth, New Jersey
  - Ocean City, New Jersey
  - New York, New York
  - VA Medical Center, Syracuse, New York
  - Upstate Gastroenterology Associates, PC, Troy, New York
  - LeBauer Research Associates, PA, Greensboro, North Carolina
  - Bethany Medical Center, High Point, North Carolina
  - Boice-Willis Clinic, Rocky Mount, North Carolina
  - Consultants for Clinical Research, Inc., Cincinnati, Ohio
  - Avamar Center for Gastroenterology, Inc., Warren, Ohio
  - Charleston Gastroenterology Specialists, LLC, Charleston, South Carolina
  - Hillcrest Clinical Research LLC, Simpsonville, South Carolina
  - Gastroenterology Associates, Kingsport, Tennessee
  - Gastrointestinal Associates, Knoxville, Tennessee
  - Memphis Gastroenterology Group, Memphis, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Clinical Trial Network, Houston, Texas
  - NationsMed Clinical Research, Houston, Texas
  - Houston Digestive Disease Clinic, Houston, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Seattle Gastroenterology Associates, Seattle, Washington
  - Eastern Washington Clinical Research Center, Spokane, Washington
  - Spokane Digestive Disease Center Research, Spokane, Washington
  - Tacoma Digestive Disease Research Center, Tacoma, Washington